CLINICAL TRIAL: NCT07066033
Title: Getting Into the Guts of Eating Disorders in Children and Adolescents. A Perspective From Psychoneuroimmunology.
Brief Title: A Study of the Intestinal Microbiota in Children and Adolescents With Eating Disorders. A Perspective From Psychoneuroimmunology
Acronym: PSYNIGED
Status: Recruiting | Type: Observational
Sponsor: Esther Nova (Other Government)
Collaborators: Spanish National Research Council (ICTAN, CSIC) (Unknown); FUNDACION PARA LA INVESTIGACIÓN BIOMÉDICA HOSPITAL INFANTIL UNIVERSITARIO NIÑO JESUS (Unknown)
Responsible Party: Sponsor-Investigator, Esther Nova, Principal Investigator, Spanish National Research Council
Organization: Spanish National Research Council (Other Government)
Other Study IDs: PID2022-136588OB-C21
Record Dates: First submitted 2025-06-17; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Eating Disorders in Adolescence; Eating Disorders in Children
Keywords: Eating disorders; psychopathology; intestinal microbiota; diettary pattern; neuroendocrine peptides; neurotransmitters; inflammation; short chain fatty acids; metagenomics; prognostic factors
MeSH Terms: conditions — Feeding and Eating Disorders; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and stool samples will be stored beyond the end of the project for a maximum period of five years. Pseudonymised samples may be used for further analyses of the same nature only if the volunteer has given consent for their use beyond the present project. Only the use by the same research team responsible for the present project will be allowed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eating disorder patients: Children and adolescents with a recent onset eating disorder initiating treatment in a Specialized Eating Disorder Unit
- Control group: Healthy children and adolescents matched by age and sex with the ED patients

SUMMARY:
The goal of this observational study is to learn if behavioral and psychological factors are associated with the intestinal microbiota composition and function in children and adolescents with eating disorders (ED). The main questions it aims to answer are:

* Are there any differences between the microbiota composition and function in adolescent patients with eating disorders and healthy adolescents?
* Are the dietary pattern and other lifestyle habits associated with the intestinal microbiota composition in patients with a recent onset eating disorder?
* Is it possible to predict the treatment response at one year by looking at any of the psychological and biological factors measured in the patients at baseline?
* Are there any differences in the intestinal microbiota among patients with different subtypes of anorexia nervosa (restrictive, binge-purging, atypical) or with avoidance/restrictive food intake disorder (ARFID)? Researchers will compare the results with those obtained from a group of healthy children and adolescents matched by sex and age to find out if the associations observed differ between ED and control participants.

Participants with ED will fill in different lifestyle questionnaires and psychological tests; they will also undergo anthropometrical measurements and will provide fecal and blood samples at baseline and one year later. Healthy participants will provide the same lifestyle information, anthopometrical measurements and stool and blood samples. They will only undergo the baseline evaluation.

DETAILED DESCRIPTION:
BACKGROUND: Eating disorders (ED) are severe and complex psychiatric pathologies characterised by the presence of abnormal eating patterns. There is not an easy cure, the clinical courses are long and often present medical, psychiatric and family complications that influence their evolution and prognosis. Almost half of the patients continue with symptoms many years after their first episode. So far, the etiology of AN remains unclear but it certainly seems to encompass multiple intertwined genetic and environmental factors, that seem to affect appetite, behavioral pathways, psychological traits and hypothalamic-pituitary-adrenal (HPA) axis dysregulation. Socio-cultural and familiar factors may favor the onset of an ED. More specifically, there are hypotheses involving brain neurotransmitters and dysregulation of reward systems, via pathways in which the gut-brain axis may be involved. The gut microbiota synthesizes or regulates the production of short-chain fatty acids (SCFAs), bile acids, tryptophan metabolites, and various neurotransmitters and hormones that may affect the central nervous system.

AIM: the study investigates whether the composition and function of the intestinal microbiota in children and adolescents with eating disorders are different from those of healthy children and adolescents. Secondarily, the relationship between the dietary pattern prior to enrollment, the psychopathology symptoms and the intestinal microbiota will be assessed.

STUDY DESIGN: a cross-sectional controlled study will be performed where the microbiota of children and adolescents with ED (AN any subtype or ARFID) will be compared with that of healthy participants matched by sex and age.

SUBJECTS: All patients referred to the specialized ED unit of the Hospital Infantil Universitario Niño Jesús that fulfill inclusion and exclusion criteria and who are willing to participate will be included. Diagnosis will be performed by psychiatrists with DSM-5 criteria.

The following information will be gathered during the interview: i) developmental history, ii) medical and psychiatric history, iii) Behaviors around the ED, iv) psychopharmacological treatment, v) sleep quality and quantity.

Healthy children and adolescents matched by sex and age will be included used as control group, who will be enrolled at their education centers.

BIOMARKER ANALYSES:

1. anthropometry and body composition study (BMI Z-score, arm circumference and tricipital skinfold thickness, bioimpedance analysis)
2. blood biomarkers: hematology, routine biochemistry, insulin, cortisol, T3; Leptin, active Ghrelin, Total PYY, active GLP-1, adiponectin, plasma inflammatory cytokines, intestinal permeability mediators of inflammation and neurotransmitters.
3. fecal biomarkers: intestinal microbiota composition analysis using shot-gun metagenomic and deep sequencing and functional genetic mechanisms; neurotransmitters (HPLC), short-chain fatty acids.

PSYCHOMETRIC TESTS: aiming the assessment of i) ED specific psychopathology (EDI-II) ii) comorbidities (anxiety and depression), iii) personality, iv) stressful life events. The family will also fill in i) ED symptoms, ii) care giver experience, iii) parental functioning.

DIETARY STUDY: includes i) 24-hour recall, ii) food frequency questionnaire over the last 15 days and iii) questionnaire on dietary habits. Dietary patterns and diet quality indexes will be derived.

STOOL PROCESSING: Stool samples, at least the size of a walnut are stored at -80C until different aliquots are separated and weighed into processing tubes for the different techniques. For fecal microbiota composition analysis specimens are analyzed as follows: bacterial DNA extraction with chromatographic column and a prior optimization step, shot-gun Illumina DNA sequencing, generation of Operational Taxonomic Unit (OTU) tables at different taxonomic levels, functional gene annotation. The DNA purification is done at the Institute of Food Science, Technology and Nutrition, CSIC and the shot-gun sequencing and bioinformatic analysis at the Microbiological Unit of the Hospital Ramón y Cajal, Madrid, Spain.

SAMPLE SIZE: previous data on microbiota in the pediatric population with ED are lacking as well as those of healthy children from the reference population. The sample size calculation performed was based on an expected effect of moderate-large size according to published findings comparing AN patients and healthy women microbiota and SCFA. For the current study to prove a medium effect size (d=0.45) in the microbiota variables with a confidence level 95% and power 80%, the result was 79 subjects per group. The ex-post power of the differences observed will be calculated.

STATISTICAL METHODS: To identify significant and predictive factors among psychological, clinical and biological variables studied, multivariate predictive models will be run on the different outcomes: binary and multidimensional. The predictive models will be chosen according to the statistical restrictions of the data.

ONE YEAR FOLLOW UP ASSESSMENT: one year after entering the study, participating patients, only, will be evaluated with the same procedures as in the baseline study to check the differences in microbiota composition with time and study potentially prognostic factors.

ETHICS: The study is approved by the Research Ethics Committee at the Hospital Infantil Universitario Niño Jesús (reference number: 0068/23. 28 November 2023) and the Ethics Committee at the Spanish National Research Council (CSIC) (reference number: 245/2023. 22 January 2024). All sensitive information of personal or biological origin will be treated with confidentiality and according to the Spanish law. All biological specimens will be treated according to specified storage, reutilization and discarding procedures as consented by the participating subjects or their legal representatives.

PERSPECTIVES: The results and findings derived from this study will help understand whether the intestinal microbiota contributes to AN etiopathology and might provide evidence to support treatment strategies for personalized treatments and better disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 7-17.9 years
* Diagnosis of Anorexia Nervosa, both restrictive (ANR) and binge-purging (ANBP) subtypes, Other Specified Feeding and Eating Disorders (OSFED), Avoidant/Restrictive Food Intake Disorder (ARFID) according to DSM-V (APA, 2013).
* Males and females
* First episode or less than 1 year evolution since initial symptoms
* Written informed consent by parent/tutor and also by the adolescent if age is more than 12 y.

Exclusion Criteria:

* Comorbidities: Current infectious disease at admission; Severe neurodevelopmental disorders with impaired language development; Moderate or severe intellectual disability; Endocrine disorders such as diabetes mellitus or thyroid disease; Celiac disease; Suicidal behaviors in the previous 3 months.
* Patients with previous unsuccessful treatments for more than one year.
* Use of the following medications before entering the study: laxatives, anabolic steroids, immunosuppressant drugs, Helicobacter pylori eradication treatment, thyroid hormones or antibiotic treatment in the previous two months
* Surgery in the previous month. Control group participants' exclusion criteria are the same plus the following: History with diagnosis of mental disease (including EDs). Current autoimmune or infectious disease.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients will be recruited in the ED specialized unit of the Niño Jesus University Children Hospital (NJUCH) after receiving a DSM-V ED diagnosis by an experienced psychiatrist. Patients will be eligible on treatment modalities including hospitalization, outpatient consultations or home hospitalization.
  The control group will be recruited among healthy children and adolescents attending eligible levels in private and public centers of formal education. Eligible educational centers are those located in geographical areas included in the administrative health zones assigned to the NJUCH. A combination of private and public schools from both metropolitan and peripheral cities is being selected. Invitation letters are sent to the head of the schools and following acceptance, randomization of age levels across schools is performed.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiota composition | Baseline
  Intestinal microbiota composition as derived from Shot-gun metagenomics with deep-sequencing analysis will be used on stool isolated DNA.
Intestinal microbiota function | Baseline
  Microbial metabolites will be analyzed in fecal water, including SCFA by gas chromatography-FID and aminoacids and neurotransmitters (GABA, dopamine, serotonin) by HPLC.

SECONDARY OUTCOMES:
Hematology | baseline
  White blood cells (WBC) and differential.
Routine biochemistry | Baseline
  Glucose, hepatic enzymes (GOT, GPT, gamma-GT), urea, creatinine, uric acid, total bilirubin; C-reactive protein, lipid profile (Cholesterol, HDL-cho, LDL-cho, VLDL-cho).
Hormones, gastrointestinal and adipose tissue peptides | Baseline
  Insulin, Cortisol, Leptin, active Ghrelin, Total PYY, active GLP-1; and Adiponectin.
Systemic Inflammation | Baseline
  plasma inflammatory cytokines (MCP-1, IL-2; IL-1beta, IL-6, TNF-alfa; IL-10); markers of intestinal permeability mediators of inflammation, such as LPS-binding protein (LPB) and zonulin-1.

OTHER OUTCOMES:
Change from baseline in fecal microbial taxa quantified by shotgun metagenomics with deep sequencing analysis | Baseline and 12 months
  In participating patients a second stool sample with be collected after one year of treatment in order to compare data on microbiota composition with baseline results.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Nova, PhD, Study Chair — Spanish National Research Council (CSIC - ICTAN); Mar Faya, PhD, MD, Principal Investigator — Hospital Infantil Universitario Niño Jesús
Locations (2):
- Spain (2):
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid
  - Institute of Food Science and Technology and Nutrition (ICTAN, CSIC), Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
* Dataset (xls or csv format) with pseudanonymization including: demographic and socioeconomic variables, diagnostic data, blood and fecal biomarkers, body composition parameters, symptoms and psychological test scores.
  * Metagenomic sequencing FASTQ files obtained from human fecal samples
Supporting Information: Study Protocol
Time Frame: Beginning after publication with no end date